CLINICAL TRIAL: NCT03321708
Title: Respiratory Microbiome in COPD. Relationship With Systemic and Pulmonary Inmune Response.
Brief Title: Respiratory Microbiome in COPD and Associated Inmune Response.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MIC-2015-57
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease (COPD), Chronic Obstructive
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, oral swabs, oral lavage, saliva, brochoalveolar lavage (BAL), bronchial brush, peripheral blood, feces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis:

COPD patients with frequent exacerbations have different pulmonary and systemic immune response than COPD patients without frequent exacerbations and this is related to their microbiome.

DETAILED DESCRIPTION:
The objective of this project is to determine the pulmonary microbiome and its relationship with the pulmonary and systemic inmune response in COPD patients with frequent (FE) and non frequent exacerbations (NE).

1. The pulmonary immune response.

   -The role of mucins, antimicrobial peptides (AMPs), Matrix metalloproteinases (MMPs) and Toll-like receptors (TLRs) as lung defense mechanisms and their possible relationship with the microbiome in COPD and FE patients.
2. The systemic immune response. -The pulmonary and blood inflammatory response and circulating bacterial products as markers of the systemic immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD according to national and international guidelines.
2. Clinical stability (8 previous weeks).
3. Signature of informed consent.

Exclusion Criteria:

1. Antibiotic treatment the previous 8 weeks.
2. Other lung diseases.
3. Active neoplasic disease.
4. Terminal concomitant disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinically stable COPD patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Relationship of pulmonary microbiome with the immune response (local and systemic). | 6 months
  Microbiome will be determined by using 16s RNA techniques. The inmune response will be studied with ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Sibila Vidal, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Oriol Sibila Vidal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mizgerd JP. Respiratory infection and the impact of pulmonary immunity on lung health and disease. Am J Respir Crit Care Med. 2012 Nov 1;186(9):824-9. doi: 10.1164/rccm.201206-1063PP. Epub 2012 Jul 12. PMID 22798317
- [Background] Roy MG, Livraghi-Butrico A, Fletcher AA, McElwee MM, Evans SE, Boerner RM, Alexander SN, Bellinghausen LK, Song AS, Petrova YM, Tuvim MJ, Adachi R, Romo I, Bordt AS, Bowden MG, Sisson JH, Woodruff PG, Thornton DJ, Rousseau K, De la Garza MM, Moghaddam SJ, Karmouty-Quintana H, Blackburn MR, Drouin SM, Davis CW, Terrell KA, Grubb BR, O'Neal WK, Flores SC, Cota-Gomez A, Lozupone CA, Donnelly JM, Watson AM, Hennessy CE, Keith RC, Yang IV, Barthel L, Henson PM, Janssen WJ, Schwartz DA, Boucher RC, Dickey BF, Evans CM. Muc5b is required for airway defence. Nature. 2014 Jan 16;505(7483):412-6. doi: 10.1038/nature12807. Epub 2013 Dec 8. PMID 24317696
- [Background] Kirkham S, Kolsum U, Rousseau K, Singh D, Vestbo J, Thornton DJ. MUC5B is the major mucin in the gel phase of sputum in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Nov 15;178(10):1033-9. doi: 10.1164/rccm.200803-391OC. Epub 2008 Sep 5. PMID 18776153
- [Background] Fujisawa T, Chang MM, Velichko S, Thai P, Hung LY, Huang F, Phuong N, Chen Y, Wu R. NF-kappaB mediates IL-1beta- and IL-17A-induced MUC5B expression in airway epithelial cells. Am J Respir Cell Mol Biol. 2011 Aug;45(2):246-52. doi: 10.1165/rcmb.2009-0313OC. Epub 2010 Oct 8. PMID 20935193
- [Background] Yang D, Biragyn A, Hoover DM, Lubkowski J, Oppenheim JJ. Multiple roles of antimicrobial defensins, cathelicidins, and eosinophil-derived neurotoxin in host defense. Annu Rev Immunol. 2004;22:181-215. doi: 10.1146/annurev.immunol.22.012703.104603. PMID 15032578
- [Background] Harder J, Meyer-Hoffert U, Teran LM, Schwichtenberg L, Bartels J, Maune S, Schroder JM. Mucoid Pseudomonas aeruginosa, TNF-alpha, and IL-1beta, but not IL-6, induce human beta-defensin-2 in respiratory epithelia. Am J Respir Cell Mol Biol. 2000 Jun;22(6):714-21. doi: 10.1165/ajrcmb.22.6.4023. PMID 10837369
- [Background] Parameswaran GI, Sethi S, Murphy TF. Effects of bacterial infection on airway antimicrobial peptides and proteins in COPD. Chest. 2011 Sep;140(3):611-617. doi: 10.1378/chest.10-2760. Epub 2011 Feb 24. PMID 21349930
- [Background] Millares L, Marin A, Garcia-Aymerich J, Sauleda J, Belda J, Monso E; PAC-COPD Study Group. Specific IgA and metalloproteinase activity in bronchial secretions from stable chronic obstructive pulmonary disease patients colonized by Haemophilus influenzae. Respir Res. 2012 Dec 11;13(1):113. doi: 10.1186/1465-9921-13-113. PMID 23228114
- [Background] Medzhitov R. Toll-like receptors and innate immunity. Nat Rev Immunol. 2001 Nov;1(2):135-45. doi: 10.1038/35100529. PMID 11905821
- [Background] Clarke TB, Davis KM, Lysenko ES, Zhou AY, Yu Y, Weiser JN. Recognition of peptidoglycan from the microbiota by Nod1 enhances systemic innate immunity. Nat Med. 2010 Feb;16(2):228-31. doi: 10.1038/nm.2087. Epub 2010 Jan 17. PMID 20081863